CLINICAL TRIAL: NCT06428695
Title: Implementation of Education on Calorie Tracking Application to Improve Adherence to a Calorie Restricted Weight Management Program
Brief Title: Education Session to Improve Program Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00110851
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-05

CONDITIONS: Weight Management
Keywords: calorie tracking; weight loss; weight management program; food intake
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: The subject population will consist of adults 18 years of age and older with a Body Mass Index (BMI) greater than 25 kg/m2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dietary self-monitoring tool education session (Experimental): access the impact of a one-hour dietary self-monitoring tool education session for participants in a calorie-restricted weight management program on their knowledge of the use of the tool to help them adhere to a calorie-restricted weight management program
  Interventions: Behavioral: one-hour dietary self-monitoring tool education session

INTERVENTIONS:
Behavioral: one-hour dietary self-monitoring tool education session — access the impact of a one-hour dietary self-monitoring tool education session for participants in a calorie-restricted weight management program on their knowledge of the use of the tool to help them adhere to a calorie-restricted weight management program
  Other Names: education session

SUMMARY:
To examine is user knowledge of a dietary self-monitoring (DSM) calorie tracking app and improving patient adherence to daily caloric food intake to help with weight loss.

DETAILED DESCRIPTION:
The research question guiding this project is: In adults with a BMI greater than 25 kg/m2, does a 1-hour education session on using a calorie-tracking application improve adherence to a calorie-restricted weight management program over eight weeks? This project aimed to increase patient knowledge with the DSM tool. To Increase adherence to the calorie-restricted diet program and, finally, to increase weight loss in the program participants of the 8-week program

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older with a Body Mass Index (BMI) greater than 25 kg/m2

Exclusion Criteria:

* Younger than18 years of age with a Body Mass Index (BMI) less than 25 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Perceived Competence Scale (PCS) Score | Baseline
  The Perceived Competence Scale (PCS) will be the open-access validated tool used for this project. This will be the 4 questions pretest/posttest utilized. A 1-hour education session will provide training on the use of a DSM calorie-tracking app. Following this will be an 8-week in-person weight management program focusing on a daily calorie and carb restriction and protein goal. Each item is scored from 1 to 4, where a score of 1 indicates low perceived competence and a score of 4 reflects high perceived competence. Scores are summed and then averaged for each subscale, resulting in four separate subscale means.
Perceived Competence Scale (PCS) Score | Week 8
  The Perceived Competence Scale (PCS) will be the open-access validated tool used for this project. This will be the 4 questions pretest/posttest utilized. A 1-hour education session will provide training on the use of a DSM calorie-tracking app. Following this will be an 8-week in-person weight management program focusing on a daily calorie and carb restriction and protein goal. Each item is scored from 1 to 4, where a score of 1 indicates low perceived competence and a score of 4 reflects high perceived competence. Scores are summed and then averaged for each subscale, resulting in four separate subscale means.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Smith, DO, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT06428695/ICF_000.pdf